CLINICAL TRIAL: NCT00218751
Title: Promoting Child Mental Health: RCT of Home Visiting
Brief Title: Early Home Visitation Program to Promote Good Health and Development in Children at Risk for Abuse
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01MH060733 (NIH); R01MH060733 (NIH); DSIR CT-P
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2008-02

CONDITIONS: Child Abuse
Keywords: Child abuse; Neglect; Home Visitation; Program Evaluation
MeSH Terms: interventions — House Calls

INTERVENTIONS:
Behavioral: Home Visiting

SUMMARY:
This study will evaluate the effectiveness of Hawaii's Healthy Start Program (HSP), a home visitation program for families at risk for child abuse, in promoting the health and development of children.

DETAILED DESCRIPTION:
Hawaii's Healthy Start Program (HSP) is a well-respected home visiting program for families at risk for abuse of their newborn children. The program incorporates early identification of at-risk families. Each family then begins receiving long-term home visitations. The home visiting component aims to promote child health and development and to prevent child abuse by improving family functioning and parenting. Home visitors are trained paraprofessionals working under professional supervision. The program includes both direct services and referrals to community resources. Direct services include providing emotional support to parents, encouraging them to seek needed professional help, teaching parents about child development, and role-modeling parenting skills and problem-solving techniques. In a previous study, at-risk families were randomly assigned to either HSP or no intervention. Evaluations were conducted at the time of the child's birth and at ages 1, 2, and 3 in order to assess the home environment and the development and well-being of the child. This study is a continuation study. Participants will include the original families from the previous study, as well as a new group of families who are not at risk for child abuse. By interviewing and observing these two groups of families, this study will evaluate the effectiveness of HSP in promoting children's mental health, cognitive and social-emotional development, and academic achievement in the first years of school.

All families will be evaluated on a yearly basis when the child is in 1st, 2nd, and 3rd grade. Interviews will be conducted with the parents, children, and teachers. Parent interviews will focus on family functioning, including mental health of the parents, parenting attitudes and behaviors, quality of the home environment, and any domestic violence or substance abuse that occurred. In addition, the child's health and development, as well as use of any community resources will be assessed. Interviews with the children and teachers will focus on assessing the child's behavior and emotional well-being. The family's home environment, the interaction between the parents and children, and the children's classroom behavior will be observed. Each child will also undergo developmental testing. All measurements will be collected at each yearly visit.

ELIGIBILITY:
Inclusion Criteria:

* Families in the Oahu community who delivered newborns between November 1994 and November 1995
* If enrolled in the control group, must not have been previously enrolled in Hawaii's Healthy Start Program

Exclusion Criteria:

* Insufficient understanding of English

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1122
Dates: Start 2000-03; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Child cognitive development, behavior, and health | At-risk sample: Up to 8 years; Not-at risk sample: Up to 2 years
Child social-emotional development | At-risk sample: Up to 6 years; Not-at risk sample: Up to 1 year
Child depression | At-risk sample: Up to 8 years; Not-at risk sample: Up to 2 years

SECONDARY OUTCOMES:
Family functioning | At-risk sample: Up to 8 years; Not-at risk sample: Up to 2 years
Parent functioning and stress levels | At-risk sample: Up to 8 years; Not-at risk sample: Up to 2 years
Substantiated reports of child abuse | At-risk sample: Up to 8 years; Not-at risk sample: Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne K. Duggan, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Duggan A, Windham A, McFarlane E, Fuddy L, Rohde C, Buchbinder S, Sia C. Hawaii's healthy start program of home visiting for at-risk families: evaluation of family identification, family engagement, and service delivery. Pediatrics. 2000 Jan;105(1 Pt 3):250-9. PMID 10617732
- [Background] Duggan A, Fuddy L, McFarlane E, Burrell L, Windham A, Higman S, Sia C. Evaluating a statewide home visiting program to prevent child abuse in at-risk families of newborns: fathers' participation and outcomes. Child Maltreat. 2004 Feb;9(1):3-17. doi: 10.1177/1077559503261336. PMID 14870994
- [Background] Duggan A, McFarlane E, Fuddy L, Burrell L, Higman SM, Windham A, Sia C. Randomized trial of a statewide home visiting program: impact in preventing child abuse and neglect. Child Abuse Negl. 2004 Jun;28(6):597-622. doi: 10.1016/j.chiabu.2003.08.007. PMID 15193851
- [Background] Duggan A, Fuddy L, Burrell L, Higman SM, McFarlane E, Windham A, Sia C. Randomized trial of a statewide home visiting program to prevent child abuse: impact in reducing parental risk factors. Child Abuse Negl. 2004 Jun;28(6):623-43. doi: 10.1016/j.chiabu.2003.08.008. PMID 15193852
- [Background] Windham AM, Rosenberg L, Fuddy L, McFarlane E, Sia C, Duggan AK. Risk of mother-reported child abuse in the first 3 years of life. Child Abuse Negl. 2004 Jun;28(6):645-67. doi: 10.1016/j.chiabu.2004.01.003. PMID 15193853
- [Background] El-Kamary SS, Higman SM, Fuddy L, McFarlane E, Sia C, Duggan AK. Hawaii's healthy start home visiting program: determinants and impact of rapid repeat birth. Pediatrics. 2004 Sep;114(3):e317-26. doi: 10.1542/peds.2004-0618. PMID 15342892
- [Background] Nelson CS, Higman SM, Sia C, McFarlane E, Fuddy L, Duggan AK. Medical homes for at-risk children: parental reports of clinician-parent relationships, anticipatory guidance, and behavior changes. Pediatrics. 2005 Jan;115(1):48-56. doi: 10.1542/peds.2004-1193. PMID 15629981
- [Background] King TM, Rosenberg LA, Fuddy L, McFarlane E, Sia C, Duggan AK. Prevalence and early identification of language delays among at-risk three year olds. J Dev Behav Pediatr. 2005 Aug;26(4):293-303. doi: 10.1097/00004703-200508000-00006. PMID 16100502
- [Background] Stone KE, Burrell L, Higman SM, McFarlane E, Fuddy L, Sia C, Duggan AK. Agreement of injury reporting between primary care medical record and maternal interview for children aged 0-3 years: implications for research and clinical care. Ambul Pediatr. 2006 Mar-Apr;6(2):91-5. doi: 10.1016/j.ambp.2005.10.003. PMID 16530145
- [Background] Duggan AK, McFarlane EC, Windham AM, Rohde CA, Salkever DS, Fuddy L, Rosenberg LA, Buchbinder SB, Sia CC. Evaluation of Hawaii's Healthy Start Program. Future Child. 1999 Spring-Summer;9(1):66-90; discussion 177-8. PMID 10414011
- [Background] Bair-Merritt MH, Jennings JM, Chen R, Burrell L, McFarlane E, Fuddy L, Duggan AK. Reducing maternal intimate partner violence after the birth of a child: a randomized controlled trial of the Hawaii Healthy Start Home Visitation Program. Arch Pediatr Adolesc Med. 2010 Jan;164(1):16-23. doi: 10.1001/archpediatrics.2009.237. PMID 20048237
- [Background] McFarlane E, Dodge RA, Burrell L, Crowne S, Cheng TL, Duggan AK. The importance of early parenting in at-risk families and children's social-emotional adaptation to school. Acad Pediatr. 2010 Sep-Oct;10(5):330-7. doi: 10.1016/j.acap.2010.06.011. PMID 20816655
- [Background] Crowne SS, Juon HS, Ensminger M, Burrell L, McFarlane E, Duggan A. Concurrent and long-term impact of intimate partner violence on employment stability. J Interpers Violence. 2011 Apr;26(6):1282-304. doi: 10.1177/0886260510368160. Epub 2010 Jun 28. PMID 20587457
- [Background] Crowne SS, Gonsalves K, Burrell L, McFarlane E, Duggan A. Relationship between birth spacing, child maltreatment, and child behavior and development outcomes among at-risk families. Matern Child Health J. 2012 Oct;16(7):1413-20. doi: 10.1007/s10995-011-0909-3. PMID 22057656
- [Background] Bair-Merritt MH, Ghazarian SR, Burrell L, Duggan A. Patterns of Intimate Partner Violence in Mothers At-Risk for Child Maltreatment. J Fam Violence. 2012 May 1;27(4):287-294. doi: 10.1007/s10896-012-9431-7. Epub 2012 Mar 23. PMID 22942558
- [Background] McFarlane E, Burrell L, Crowne S, Cluxton-Keller F, Fuddy L, Leaf PJ, Duggan A. Maternal relationship security as a moderator of home visiting impacts on maternal psychosocial functioning. Prev Sci. 2013 Feb;14(1):25-39. doi: 10.1007/s11121-012-0297-y. PMID 23104075